CLINICAL TRIAL: NCT05123040
Title: Ruxolitinib, Human Chorionic Gonadotropin (uhCG/EGF), and Dose De-escalated Corticosteroids for Treatment of Minnesota High-Risk Acute GVHD (aGVHD): A Phase I/II Study
Brief Title: Ruxolitinib, Human Chorionic Gonadotropin (uhCG/EGF), and Dose De-escalated Corticosteroids
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020LS098; MT2020-28 (Other: Masonic Cancer Center)
Record Dates: First submitted 2021-11-03; First posted 2021-11-17 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Acute-graft-versus-host Disease
Keywords: aGVHD
MeSH Terms: interventions — ruxolitinib; Chorionic Gonadotropin; Adrenal Cortex Hormones; Prednisone; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ruxolitinib;hCG (Pregnyl®) ;Corticosteroids (Experimental): * Ruxolitinib 10 mg by mouth twice daily (with dose adjustments as indicated) through day 56, followed by taper
  * hCG (Pregnyl®) 2,000 units/m2 SQ every other day x 3 doses, followed by twice weekly x 14 doses (total 17 doses through day 56)
  * Corticosteroids (Prednisone, or IV methylprednisolone equivalent)
    * Dose level 1 (starting dose) = 1 mg/kg
    * Dose level 2 = 0.5 mg/kg
    * Dose level 3 = 0.25 mg/kg
    * Dose level 4 = 0.1 mg/kg
    * Dose level 5 = 0 mg/kg
  Interventions: Drug: Ruxolitinib 10 MG Oral Tablet; Drug: hCG; Drug: Corticosteroids

INTERVENTIONS:
Drug: Ruxolitinib 10 MG Oral Tablet — By mouth twice daily through day 56, then tapered
Drug: hCG — 2,000 units/m2 SQ every other day x 3 doses, followed by twice weekly x 14 doses
  Other Names: Pregnyl
Drug: Corticosteroids — Dose level 1 (starting dose) = 1 mg/kg
  * Dose level 2 = 0.5 mg/kg
  * Dose level 3 = 0.25 mg/kg
  * Dose level 4 = 0.1 mg/kg
  * Dose level 5 = 0 mg/kg
    • If dose level 1 is determined to be below the Recommended Phase 2 Dose (RP2D), the dose will be escalated:
  * Dose level -1 = 1.5 mg/kg
  * Dose level -2 = 2 mg/kg
  Other Names: Prednisone; IV methylprednisolone

SUMMARY:
This multi-center center phase I/II study to establish the lowest possible recommended phase 2 dose (RP2D) of corticosteroids in conjunction with ruxolitinib and uhCG/EGF (a novel combination) for high-risk aGVHD.

This is a single arm study designed to determine the lowest dose of corticosteroids required (toxicity endpoint) without impairing GVHD complete response or partial response (CR/PR) at day 28 when given in conjunction with uhCG/EGF and ruxolitinib.

After completion of the corticosteroid dose finding, the final dose will be carried forward into a two-stage phase II extension trial to confirm safety and make a preliminary determination of efficacy of this novel drug combination for high-risk aGVHD.

ELIGIBILITY:
Inclusion Criteria:

HCT recipients over 12 years of age within the first 7 days of initial treatment of high-risk aGVHD, defined as:

* Newly diagnosed Minnesota high-risk aGVHD -OR-
* Newly diagnosed Minnesota standard risk aGVHD with plasma amphiregulin ≥ 33 pg/ml tested at the UMN Cytokine Reference Lab. For amphiregulin lab ordering information, see Fairview Lab Guide: http://labguide.fairview.org/showtest.asp?testid=6766&format=long -OR-
* Newly diagnosed Minnesota standard risk aGVHD Ann Arbor 3 biomarkers tested by Viracor. For ordering information, see: https://www.viracor-eurofins.com/test-menu/403572p-agvhd-symptomatic- onset-algorithm/

  * Renal: Serum creatinine ≤2.5x upper limit of normal (ULN)
  * Cardiac: Left ventricular ejection fraction (LVEF) ≥ 35%
  * Voluntary written consent (adult or parent/guardian with minor assent for 12 through 17-year-olds).

Exclusion Criteria:

* Progressive malignancy
* Uncontrolled bacterial, fungal, parasitic, or viral infection at initiation of protocol treatment
* Unwilling or unable to stop supplemental sex hormone therapy (estrogen, progesterone, and/or testosterone preparations)
* Unwilling or unable to stop GnRH antagonists, aromatase inhibitors, or anti-androgens
* History of a hormone responsive malignancy
* Current thromboembolic disease requiring full-dose anticoagulation - patients receiving pharmacologic prophylaxis for thromboembolic disease will be eligible
* Active or recent (within prior 3 months) thrombus, irrespective of anticoagulation status
* Pregnancy
* Women or men of childbearing potential unwilling to take adequate precautions to avoid unintended pregnancy from the start of protocol treatment through 30 days after the last treatment

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2023-06-05 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Recommend the lowest possible dose for Phase II of corticosteroids when given in combination with ruxolitinib and uhCG/EGF in pediatric based on DLT frequency | 28 days after therapy
  Plan report patients proportions and their 95% confidence intervals of paitents who experience dose limiting toxicity. Determine best dose based on DLT criteria by CTCAE v5.0
  * Thrombosis requiring anticoagulation
  * Ascites (grade 3-5)
  * Ovarian hyperstimulation syndrome
Best response of treatment in adult and children | 28 days after therapy
  proportions of complete, partial, mixed, and no response among surviving patients at days 28 after initiation of protocol therapy in pediatric and adult patients with Minnesota high-risk aGVHD

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 30 days after treatment
  Report any type of adverse event caused by a drug cause by dose of steroids in combination of ruxolitinib and uhCG/EGF.
  Due to the complex medical condition of the GVHD patient, monitoring for adverse events will focus on the following events beginning with the date consent is signed and continuing for 30 days after the subject has completed or discontinued from the study or has taken last dose of the study drug.
  * Rehospitalization
  * Death
  * Hematologic (grade 3-5 cytopenia)
  * Infections (grade 3-5)
  * Hyperglycemia (grade 3-5)
  * Steroid myopathy (grade 3-5)
Incidence of acute GVHD flare after CR/PR requiring increase of steroids or other systemic treatment | 28 days after treatment
  Find proportion of incidence of acute GVHD
Incidence of acute GVHD flare after CR/PR requiring increase of steroids or other systemic treatment | 56 days after treatment
  Find proportion of incidence of acute GVHD
Compare the rate of treatment failure for acute GVHD after initiation of protocol therapy to historical controls | 28 days after treatment
  Compare count of treatment failure to other number of failures in other historical protocols
Compare the rate of treatment failure for acute GVHD after initiation of protocol therapy to historical controls | 56 days after treatment
  Compare count of treatment failure to other number of failures in other historical protocols
To assess patient quality of life on study | 6 month after treatment
  Have participants take an overall survival survey
Determine 1-year overall survival | 1 year post treatment
  Provide proportions and their 95% confidence intervals of patients still alive at one year post-treatment
Non-relapse mortality (death without recurrent or progressive disease after allo-HSCT) | 1 year post treatment
  Provide proportions and their 95% confidence intervals of patients who expedience a non-relapse mortality.
Collect blood samples and rectosigmoid biopsies for future correlative studies | 1 year after treament
  Give a count of the number of patients who had blood and rectosigmoid biopsies

CONTACTS AND LOCATIONS:
Overall Officials: Sherman Holtan, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota, United States